CLINICAL TRIAL: NCT03232411
Title: Biobank for African American Prostate Cancer Research in Florida
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: James and Esther King Biomedical Research Program (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-18643
Record Dates: First submitted 2017-07-17; First posted 2017-07-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: prostate disease; prostatic neoplasm; biobank; prostate cancer in black males; biospecimen; smoking and the aggressiveness of prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases; Smoking | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva samples and tumor tissue samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — Participants will be asked to complete a baseline questionnaire that asks questions about their demographic information, medical history, and smoking habits when they first enroll in the study. They will also be asked to complete a follow-up questionnaire 2 years later. The questionnaires will each take about 25 minutes to complete.
Other: Saliva Samples — Participants will be asked to provide a saliva sample using the saliva kit that will be mailed to them. Detailed instructions for collection will be included in the saliva collection packet.
Other: Tumor Tissue — Participants will be asked for permission to obtain a sample of their tumor tissue. Participants will receive a medical release form. Once they complete it and mail it back, investigators will request a small amount of tissue collected during the participant's prostate biopsy (or during their surgery, if they had surgery) from their health care provider.

SUMMARY:
The purposes of this study are: a) to develop a statewide Biobank for prostate cancer among men of African Ancestry in Florida and; b) to examine whether smoking increases the aggressiveness of prostate cancer using several biological approaches.

Investigators plan to contact African American prostate cancer patients regarding participation. This project has 3 main components. Eligible patients may choose to participate in any or all parts of the study: Questionnaires; Saliva Samples; Tumor Tissue.

DETAILED DESCRIPTION:
This project will create the first state-wide data and biospecimen bank for men of African ancestry with prostate cancer. The sampling strategy and size of the study population ensure that the cohorts is representative, enhancing validity of studies based on this resource. In addition, there are no data on the role of smoking in African American prostate cancer. The approach to share the resource with Florida prostate cancer researchers is innovative and possible because the four annual prostate cancer symposiums organized by Moffitt has unified many Florida prostate cancer researchers who are now well connected and actively collaborating, as evidenced by publications and funded projects among participants.

ELIGIBILITY:
Inclusion Criteria:

* The initial recruitment of cases will be done with 3 mailings: the first to introduce the study to the participant from Florida Cancer Data System (FCDS) of the Florida Department of Health and ask them to complete the eligibility form and contact information update form; a second mailing to those who are determined to be eligible for the study to obtain the Informed Consent Form and the Baseline survey; and a third mailing to those who completed the survey to obtain a saliva sample and medical release form for tissue.
* Histologically biopsy confirmed, primary prostate cancer, diagnosed between January 2013 and December 2015
* African American or Black; Hispanic Black; Afro-Caribbean
* Are at least 20 years old
* Are a resident of Florida
* Additional criteria may apply

Exclusion Criteria:

* Does not meet Inclusion Criteria

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men of African Ancestry in Florida who were diagnosed with prostate cancer between January 2013 and December 2015.
Sampling Method: Non-Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Number of Complete Patient Data Records Collected at Three Years | Up to 3 years
  The study timeline is up to 3 years to collect detailed patients' data, outcome information and bio-specimens from men of African Ancestry with prostate cancer (n=6,000), diagnosed between January 2013 and December 2015.

SECONDARY OUTCOMES:
Rate of Impact of Smoking in Prostate Cancer Aggressiveness - All Participants | Up to 3 years
  Rate of prostate aggressiveness according to the smoking status (never, former, current cigarette smoker, pipe/cigar smoker only) at the time of diagnosis. This smoking status can be dichotomized into current smoker and non-smoker.
Rate of Impact of Smoking in Prostate Cancer Aggressiveness - Current Smokers | Up to 3 years
  Current smokers further will be classified according to the Pack-year which will be obtained from questionnaire.
Number of Participants with Genetic Markers for Smoking Aggressiveness | Up to 3 years
  Occurrence of genetic changes associated with smoking and aggressiveness in prostate tumor samples. Investigators selected ~200 mutations identified in 12 prostate-cancer related genes (AR, ETS, TP53, PTEN, APC, BRAF, BRCA2, ATM, KRAS, SPOP, ERG and EGFR) based upon preliminary study and literature search. Investigators will perform mutation detection on randomly selected 200 patients and determine their association with aggressiveness and smoking.
Number of Participants with Epigenetic Markers for Smoking Aggressiveness | Up to 3 years
  Occurrence of epigenetic changes associated with smoking and aggressiveness in prostate tumor samples. A customized panel of 384 CpG sites will be profiled. 384 candidate CpG sites were selected from 149 sites including 18 multiple differentially methylated regions (DMRs) identified in the preliminary study, 235 sites from previous literatures. Investigators will determine their association with aggressiveness and smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Jong Park, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE